CLINICAL TRIAL: NCT06898281
Title: Effectiveness and Safety of Intracardiac Echocardiography-Guided Catheter Ablation for Premature Ventricular Contractions Originating From the Papillary Muscles: A Randomized Controlled Trial
Brief Title: Intracardiac Echocardiography-Guided Catheter Ablation for Premature Ventricular Contractions Originating From the Papillary Muscles
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Collaborators: The Second People's Hospital of Anhui Province (Other); The First People's Hospital of Hefei (Other); Qilu Hospital of Shandong University (Other); Fujian Medical University Union Hospital (Other); Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Xu Liu, Professor, Shanghai Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ICE-PMPVC
Record Dates: First submitted 2025-03-22; First posted 2025-03-27 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-03

CONDITIONS: Premature Ventricular Contractions
Keywords: intracardiac echocardiography; papillary muscle-originating premature ventricular contractions; premature ventricular contractions
MeSH Terms: conditions — Ventricular Premature Complexes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intracardiac echocardiography (ICE)-guided catheter ablation (Experimental): Intracardiac echocardiography (ICE)-guided catheter ablation.
  Interventions: Procedure: intracardiac echocardiography (ICE)-guided catheter ablation
- Pressure-sensing catheter ablation alone (Active Comparator): Pressure-sensing catheter ablation alone.
  Interventions: Procedure: Pressure-sensing catheter ablation alone

INTERVENTIONS:
Procedure: intracardiac echocardiography (ICE)-guided catheter ablation — Intracardiac echocardiography (ICE)-guided catheter ablation.
  Arms: intracardiac echocardiography (ICE)-guided catheter ablation
Procedure: Pressure-sensing catheter ablation alone — Pressure-sensing catheter ablation alone
  Arms: Pressure-sensing catheter ablation alone

SUMMARY:
This randomized, prospective, parallel, single-blind, multicenter clinical trial investigates the efficacy and safety of intracardiac echocardiography (ICE)-guided catheter ablation versus pressure-sensing catheter ablation alone in reducing PVC recurrence among patients with confirmed papillary muscle-originating premature ventricular contractions (PVCs). Participants were randomly allocated to either the ICE-guided intervention group or the conventional ablation control group following definitive diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years.
* Diagnosed with premature ventricular contractions (PVCs) originating from the papillary muscles.
* Symptoms refractory to antiarrhythmic drug therapy.
* Patients must be capable and willing to provide written informed consent for study participation.

Exclusion Criteria:

* History of cardiac surgery or any prior cardiac interventional procedures.
* Ischemic heart disease, dilated cardiomyopathy, or hypertrophic cardiomyopathy.
* Severe hepatic or renal dysfunction:

AST/ALT >3× upper limit of normal (ULN); Serum creatinine (SCr) >3.5 mg/dl or creatinine clearance (Ccr) <30 ml/min.

* Prior ablation for papillary muscle PVCs.
* Life expectancy <1 year.
* Pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2025-03-23 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Freedom from VC recurrence | Patients were followed up at 3 months postoperatively to assess recurrence.
  Freedom from VC recurrence (defined as a ≥80% reduction in VC burden, calculated as [number of VCs per 24 hours / total number of heartbeats per 24 hours] × 100%).

SECONDARY OUTCOMES:
VC burden reduction | Patients were followed up at 3 months postoperatively to assess recurrence.
  Preoperative VC burden [%] - postoperative VC burden [%].
Total procedure time | From the start to the end of the procedure.
  Total procedure time.
Total fluoroscopy time | From the start to the end of the procedure.
  Total fluoroscopy time.
Major perioperative complications | 30 days postoperatively.
  Including cardiac tamponade, atrioventricular block, stroke, or pulmonary embolism.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, Xuhui, China